CLINICAL TRIAL: NCT01517893
Title: A Phase-II, Randomized, Placebo-controlled Trial of Simvastatin in Generalized Vitiligo
Brief Title: Clinical Trial of Simvastatin to Treat Generalized Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John Harris (Other)
Responsible Party: Sponsor-Investigator, John Harris, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UM-DERM001
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Vitiligo
Keywords: vitiligo; simvastatin
MeSH Terms: conditions — Vitiligo | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Sig: Simvastatin 40 mg, increased to 80 mg after 1 month if initial dose tolerated
  Interventions: Drug: Simvastatin
- Placebo Arm (Placebo Comparator): Sig: 40 mg PO daily for 1 month, increased to 80 mg PO daily for 5 months if low dose tolerated
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin — Sig: 40 mg PO daily for 1 month, increased to 80 mg PO daily for 5 months if low dose tolerated
  Arms: Intervention arm
Drug: Placebo — Sig: 40 mg PO daily for 1 month, increased to 80 mg PO daily for 5 months if low dose tolerated
  Arms: Placebo Arm

SUMMARY:
The investigators purpose is to initiate a phase II, randomized, placebo-controlled clinical trial to test simvastatin, an FDA-approved medication for hypercholesterolemia, as a new treatment for vitiligo. The aims of this placebo-controlled study seek to determine the safety and potential efficacy of simvastatin 80mg daily versus placebo in adult male patients with generalized vitiligo. Additionally, the investigators will collect blood to examine the effect of simvastatin on autoreactive CD8+ T cells in vitiligo patients.

DETAILED DESCRIPTION:
Vitiligo is an autoimmune disease caused by autoreactive CD8+ T lymphocytes that target melanocytes, and interferon-γ-induced CXCL10 plays an important role.1 Simvastatin inhibits interferon-γ signaling by blocking activation of STAT12 and prevented and reversed disease in our mouse model.3 A case report described a patient with vitiligo who repigmented with simvastatin.4 We conducted a small, randomized, double-blind, placebo-controlled, phase II clinical trial to test simvastatin as a treatment for vitiligo. After obtaining informed consent, we enrolled men ages 18 to 64 years with vitiligo affecting 3% to 50% of their body surface area (BSA). We excluded patients with a segmental presentation; those already taking 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitor; those with existing thyroid disease; and women, based on their increased risk of simvastatin-induced myopathy.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* ages 18-64
* at least one vitiligo skin lesion measuring at least 2x2 cm in size
* willing and able to understand and sign informed consent
* able to complete study and comply with study procedures

Exclusion Criteria:

* history of segmental vitiligo
* allergy to statin medications
* use of statin medications due to cardiac risks.
* use of any medications contraindicated with use of simvastatin
* use of topical vitiligo treatments in past 4 weeks
* use of laser or light-based vitiligo treatments within the past 8 weeks
* treatment with immunomodulating oral medications in the past 4 weeks
* use of statin medications in the past 8 weeks
* evidence of hepatic dysfunction, personal or family history of non-alcoholic steatotic hepatitis, or personal history of hepatitis
* evidence of renal dysfunction
* history of myopathy or rhabdomyolysis, or elevated baseline creatinine kinase
* recent history of alcohol or drug abuse
* history of diabetes
* untreated hypothyroidism
* other conditions that require the use of interfering topical or systemic therapy
* other current conditions that might interfere with study assessments such as, but not limited to, atopic dermatitis and psoriasis
* clinically significant abnormal findings or conditions which might, in the opinion of the Principal Investigator, interfere with study evaluations or pose a risk to subject safety during the study.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E. Harris, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School Clinical Research Center, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Placebo Arm
Started | 8 | 7
Completed | 5 | 7
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Placebo Arm | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [28 to 55] | 39 [32 to 49] | 41.6 [28 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 7 | 15
Vitiligo area scoring index [Mean (Full Range); unit: percentage] — The vitiligo area scoring index (VASI) is a measure of the surface area affected by vitiligo in a given research subject. It ranges from 0% (no vitiligo) to 100% (complete depigmentation of the entire body surface area). In terms of treatment, a decrease in VASI is desirable as it indicates less surface area affected by vitiligo. The score represents an estimate made by the investigators, based on the approximation that one "hand unit," is roughly equivalent to 1% of the body surface area.
  percentage | 14.81 [3.23 to 40.93] | 23.09 [5.12 to 46.26] | 19.23 [3.23 to 46.26]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in Vitiligo Area Scoring Index (VASI) Score
Description: Number of participants with 33% decrease in the Vitiligo Area Scoring Index (VASI) from baseline to the last available study visit.
  Decrease in VASI score means improvement. Minimum value is 0, that means no vitiligo. maximum value is 100, that means 100% of the body surface area has vitiligo (total body surface area).
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Population: Overall number of participants for intervention (5) differs from enrollment (8) due to withdraw of 3 participants on intervention arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 7
Participants | 0 | 0

2. Secondary Outcome: Number of Participants With Increase in Investigator's Global Assessment Score
Description: Increase in Investigator Global Assessment Scores of 30% or more from baseline to last available visit.
  Increase in score means improvement. 0% is no improvement at all. 100% is complete recovery.
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Population: For placebo arm, only 6 out of 7 participants reported data.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 6
Participants | 1 | 0

3. Secondary Outcome: Number of Participants Experiencing Toxicity From of High-dose Simvastatin .
Description: The number of participants who experienced toxicity based upon monitored lab values (Liver Function Test) and patient symptoms for evidence of simvastatin toxicity
Time Frame: Assessed at baseline, then monthly until final study visit, six months after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 7
Participants | 0 | 0

4. Secondary Outcome: Change in Sentinel Patch Area
Description: Change in percent depigmentation of sentinel patch lesion from baseline to last available study visit ( 6 months after randomization).
  positive numbers mean increase or worsening of sentinel patch area negative numbers mean decrease or improvement of sentinel patch area
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Measure: Mean (Standard Deviation); unit: cm2
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 7
cm2 | -0.2272 (3.463) | 3.8571 (9.17)

5. Secondary Outcome: Change in Quality of Life Score by Using DERMATOLOGY LIFE QUALITY INDEX (DLQI)
Description: The aim of this questionnaire is to measure how much your skin problem has affected your life. We measured change in questionnaire score from baseline to end of study (at 6 months after randomization) of subjects randomized to treatment with simvastatin versus placebo. Change was measured as a drop in score at the end of 6 months of treatment.
  Minimum score is 0, maximum is 30. Higher value means worse score.
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 7
units on a scale | 3.4 (4.159326869) | 2.285714286 (2.690370837)

6. Secondary Outcome: Number of Participants With an Increase in Patient's Global Assessment Score
Description: Increase in Patient's Global Assessment Scores of 30% or more from baseline to last available visit Increase means improvement. minimum is 0% and maximum is 100%
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Population: Placebo arm reports 6 instead of enrolled 7 due to failure of participant to complete assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 5 | 6
Participants | 0 | 1

7. Secondary Outcome: Serum CXCL10 Levels From the First and Last Available Clinic Visits Were Measured Via ELISA
Description: Determination of the effects of simvastatin treatment on Serum CXCL10 levels from the first and last available clinic visits were measured via ELISA in the blood of patients with vitiligo treated with simvastatin versus placebo
Time Frame: Assessed at baseline and final study visit, 6 months after randomization
Population: Serum CXCL10 levels from the first and last available clinic visits were measured via ELISA. The mean and SEM are reported here. One participant in intervention group was not included because participant withdrew before a second CXCL10 level was obtained. Other withdrawn participants were included, using the CXCL10 from their final visits.
Measure: Mean (Standard Error); unit: Fold change of baseline CXCL10 level
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 7 | 7
Fold change of baseline CXCL10 level | 0.9148 (0.263) | 0.6176 (0.1685)

8. Secondary Outcome: CXCR3 Expression on CD8+ T Cells
Description: Determination of the effects of simvastatin treatment on CXCR3 expression in melanocyte-specific, autoreactive CD8+ T cells in the blood of patients with vitiligo treated with simvastatin versus placebo
Time Frame: Assessed prior to treatment and periodically while on treatment
Population: No data collected as this outcome was abandoned due to budget constraints and strength of other study results.
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months (baseline to end of treatment)
Description: Safety lab values and questionnaires collected for outcomes.
Arm/Group | Intervention Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7
Other Adverse Events (participants affected / at risk) | 4/8 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=8) | Placebo Arm (N=7)
Burn (Skin and subcutaneous tissue disorders) | 1 | 0 — Sustained at work, unrelated
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention Arm (N=8) | Placebo Arm (N=7)
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
leg twinge (Musculoskeletal and connective tissue disorders) | 0 | 1
diarrhea (Gastrointestinal disorders) | 1 | 2
abdominal pain (Gastrointestinal disorders) | 0 | 1
tinnitus (Ear and labyrinth disorders) | 0 | 1
flatulence (Gastrointestinal disorders) | 0 | 1
stool odor (Gastrointestinal disorders) | 0 | 1
pulled muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
arthrlagia (Musculoskeletal and connective tissue disorders) | 2 | 0
URI symptoms (Respiratory, thoracic and mediastinal disorders) | 1 | 2
xerosis (Skin and subcutaneous tissue disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
urine color change (Renal and urinary disorders) | 1 | 0
sleep disturbance (Nervous system disorders) | 1 | 0
dental infection (Infections and infestations) | 1 | 0

LIMITATIONS AND CAVEATS:
The following outcome measures were abandoned: 1.Decrease in CXCR3 exp. on CD8 positive T-Cells, 2.Corr. Among Var. Outcome Measures for Vitiligo: procedures not performed/no data collected due to strength of prior outcomes & budget limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes